CLINICAL TRIAL: NCT00050661
Title: Use of Humanized CD25 (Anti-TAC) Monoclonal Antibody/ Placebo to Prevent Relapse of Psoriasis Vulgaris Following NBUVB Therapy
Brief Title: To Study the Use of Humanized CD25 in Preventing the Relapse of Psoriasis Vulgaris
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Facet Biotech (Industry)
Responsible Party: James Krueger, MD, PhD, Rockefeller University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JKR-0337
Record Dates: First submitted 2002-12-17; First posted 2002-12-18 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Psoriasis
Keywords: psoriasis; Cyclosporine; Daclizamub; anti-TAC; dermatology; skin; lesions
MeSH Terms: conditions — Psoriasis | interventions — Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narrow Band Ultraviolet B (Active Comparator): 312nm
  Interventions: Device: NB-UVB
- anti-TAC or placebo (Experimental)
  Interventions: Drug: Daclizumab

INTERVENTIONS:
Drug: Daclizumab — Humanized anti-CD25 antibodies (anti-TAC), or placebo (saline solution), will be given as intravenous infusions on the following schedule: 2 mg/kg initially (maximum dose 200 mg) infusion given over 60 minutes, followed by a 1 mg/kg (maximum of 100 mg) infusion given over 30 minutes every two weeks thereafter for a total of 8 doses.
  Other Names: anti-TAC
  Arms: anti-TAC or placebo
Device: NB-UVB — total body NB-UVB at a dose that is 50% of the MED. Patients are treated 3-7 times per week, with increasing doses at every treatment if no burning occurs. This is continued until for a total of 20 ± 2 treatments total.
  Arms: Narrow Band Ultraviolet B

SUMMARY:
This study is designed to study disease relapse after NBUVB and how the administration of Daclizumab/placebo alters disease relapse.

DETAILED DESCRIPTION:
The first part of the study involves NB-UVB light treatment, a well-established treatment to treat psoriasis. In the second part, we are testing a drug known as Humanized CD25 Monoclonal Antibody (anti-TAC) or placebo to prevent disease relapse. Anti-TAC is an injectable medicine that is also designed to treat psoriasis by blocking a part of the immune system that we believe contributes to the disease.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients with chronic psoriasis vulgaris (disease stable or worsening for > 6 months). Patients age 16 - 21 will be considered on a case to case basis.

   For those patients under the age of 18, parental consent will be obtained.
2. Extensive skin involvement.
3. Scale, thickness, and erythema in individual psoriasis lesions of at least moderate intensity.
4. Psoriasis treated with emollients only for 2 weeks prior to treatment
5. Patients with active psoriatic arthritis, if accompanied by psoriasis vulgaris involving more than 5% of the body surface.
6. Patients that are appropriate for treatment with UVB.

Exclusion Criteria:

1. Positive serology for HIV, Hepatitis B, or Hepatitis C.
2. Positive β-HCG titer. For women of childbearing potential, unwillingness or inability to use a contraceptive device during this study if negative for β-HCG.
3. Guttate psoriasis, pustular psoriasis, or whole body erythroderma.
4. Active infection or persistent fever of unknown origin.
5. Major concurrent illness, which could worsen following treatment with anti-TAC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1997-10; Primary Completion 2004-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
time to disease relapse | After a course of NB-UVB treatment

SECONDARY OUTCOMES:
Histologic assessment of disease activity at relapse for measures of epidermal hyperplasia, leukocyte infiltration, and expression of cytokine-induced inflammatory proteins. | before and after NB-UVB treatment

CONTACTS AND LOCATIONS:
Overall Officials: James Krueger, MD, PHD, Principal Investigator — Rockefeller University
Locations (2):
- United States (2):
  - Rockefeller University Hospital, New York, New York
  - Rockefeller University, New York, New York